CLINICAL TRIAL: NCT00101257
Title: Phase I Study to Evaluate the Safety of Cellular Adoptive Immunotherapy Using Autologous CD4+ Antigen-Specific T Cell Clones for Patients With Advanced Ovarian Cancer
Brief Title: Cellular Adoptive Immunotherapy in Treating Patients With Stage III or Stage IV Ovarian Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 1942.00; FHCRC-1942.00; CDR0000402870 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes

SUMMARY:
RATIONALE: Biological therapies, such as cellular adoptive immunotherapy, stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase I trial is studying the side effects and best dose of cellular adoptive immunotherapy in treating patients with stage III or stage IV ovarian cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity of autologous CD4-positive antigen-specific T cells in patients with stage III or IV ovarian epithelial cancer or primary peritoneal cavity cancer.
* Determine the duration of in vivo persistence of this drug in these patients.

Secondary

* Determine the antitumor effect of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients undergo leukapheresis for collection of T cells. Responder T cells are stimulated in vitro with autologous peripheral blood mononuclear cell-derived dendritic cells pulsed with NY-ESO-1 immunogenic peptides. Patients receive autologous CD4-positive antigen-specific T cells IV over 30 minutes.

Cohorts of 3-6 patients receive escalating doses of autologous CD4-positive antigen-specific T cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 4, 8, and 12 weeks and then periodically thereafter for survival.

PROJECTED ACCRUAL: A total of 9-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV ovarian epithelial cancer or primary peritoneal cavity cancer meeting 1 of the following criteria:

  * Progressive* or persistent* disease during or after primary chemotherapy
  * Recurrent disease < 6 months after completion of primary therapy that had resulted in a complete response
  * Persistent* or recurrent disease after second-line or additional therapies NOTE: *Progression or persistence can be based on serological (CA 125 > 100 U/mL OR 2 times baseline), radiographic (measurable or evaluable disease), or second-look surgical findings
* Tumor expressing NY-ESO-1 determined by IHC or RT-PCR
* HLA type expressing DPB*0401, DPB1*0201, DRB1*07
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 16 weeks

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No congestive heart failure*
* No clinically significant hypotension*
* No symptoms of coronary artery disease*
* No cardiac arrhythmias on EKG requiring drug therapy*
* No history of cardiovascular disease*
* No other significant cardiovascular abnormalities* NOTE: *Patients with any of the above undergo a stress test and/or echocardiography before being determined ineligible for study participation

Pulmonary

* FEV_1 ≥ 60% of predicted*
* DLCO ≥ 55%* NOTE: *Patients with clinically significant pulmonary dysfunction only

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No active infection
* No oral temperature > 38.2°C within the past 72 hours
* No systemic infection requiring chronic maintenance or suppressive therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy (e.g., interleukins, interferons, vaccines, intravenous immunoglobulin, or expanded polyclonal tumor-infiltrating lymphocytes or lymphokine-activated killer cell therapy)

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior standard or experimental chemotherapy

Endocrine therapy

* No concurrent systemic corticosteroids except for treatment-related toxicity

Radiotherapy

* At least 3 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 3 weeks since prior immunosuppressive therapy
* More than 3 weeks since prior investigational drugs and recovered
* No other concurrent investigational agents
* No concurrent pentoxifylline

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-10; Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity
Duration of in vivo persistence
Antitumor effects

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States